CLINICAL TRIAL: NCT03284853
Title: A Prospective, Double-masked, Randomized, Multicenter, Active-controlled, Parallel-group, 6-month Study Assessing the Safety and Ocular Hypotensive Efficacy of PG324 Ophthalmic Solution Compared to GANFORT® (Bimatoprost 0.03% / Timolol 0.5%) Ophthalmic Solution in Subjects With Elevated Intraocular Pressure (MERCURY 3)
Brief Title: Safety and Efficacy Study of PG324 (Netarsudil/Latanoprost 0.02% / 0.005%) Ophthalmic Solution Compared to GANFORT® Ophthalmic Solution in Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG324-CS303
Record Dates: First submitted 2017-08-29; First posted 2017-09-15 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — netarsudil; Latanoprost; Ganfort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Netarsudil/Latanoprost 0.02%/0.005% (Experimental): PG324 Ophthalmic Solution (netarsudil 0.02% / latanoprost 0.005%) one drop daily to each eye for 180 days.
  Interventions: Drug: Netarsudil/Latanoprost 0.02%/0.005%
- GANFORT® (Active Comparator): GANFORT® (bimatoprost 0.03%/timolol 0.5%) Ophthalmic solution one drop daily to each eye for 180 days.
  Interventions: Drug: GANFORT®

INTERVENTIONS:
Drug: Netarsudil/Latanoprost 0.02%/0.005% — Topical sterile ophthalmic solution
  Arms: Netarsudil/Latanoprost 0.02%/0.005%
Drug: GANFORT® — Topical sterile ophthalmic solution
  Arms: GANFORT®

SUMMARY:
The study is intended to test the effectiveness and safety of Netarsudil / Latanoprost 0.02% / 0.005% Ophthalmic Solution, relative to GANFORT® for lowering of intraocular pressure (IOP) in patients with elevated intraocular pressure

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older.
2. Diagnosis of OAG or OHT in both eyes (OAG in one eye and OHT in the fellow eye is acceptable).
3. Subjects insufficiently controlled and/or subjects considered in need for combination therapy by the investigators.
4. Medicated intraocular pressure ≥ 17 mmHg in at least one eye and < 28mmHg in both eyes at screening visit.
5. Unmedicated (post-washout) IOP >20mmHg in at least one eye and < 36mmHg in both eyes at 2 qualification visits at 08:00 hour, 2-7 days apart. At the second qualification visit, have IOP >17mmHg in at least one eye and < 36mmHg in both eyes at 10:00 and 16:00 hours. Note: For purposes of determining eligibility of subjects to be enrolled, the non-integral IOP mean number will be used. Any non-integral mean IOP number should not be rounded. If only one eye qualifies at the second qualification visit it MUST be the same eye that qualified on the first visit and this will be the study eye for the duration of the study.
6. Best corrected visual acuity +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200 or better Snellen visual acuity in each eye).
7. Be able and willing to give signed informed consent and follow study instruction.
8. Women must be either of non-childbearing potential, or women with childbearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study.
9. Women of childbearing potential must have a negative urine pregnancy test within 7 days of first dose of study treatment and agree to use highly effective contraception during the study and for 3 months after the last dose of study medication.
10. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use an effective form of contraception from time of randomization and for 3 months following the last dose of study medication.
11. In France, a subject will be eligible for inclusion in this study only if either affiliated to or as a beneficiary of a social security number.

Exclusion Criteria:

Ophthalmic:

1. Clinically significant ocular disease (e.g., corneal edema, uveitis, or severe keratoconjunctivitis sicca) which might interfere with interpretation of the study efficacy endpoints or with safety assessments, including subjects with glaucomatous damage so severe that washout of ocular hypotensive medications for 4 weeks or longer if needed is not judged safe as it would put the subject at risk for further vision loss.
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure glaucoma, or narrow angles i.e. Grade 2 Shaffer (Chan 1981) or less extreme narrow angle with complete or partial closure. Note: Previous laser peripheral iridotomy is NOT acceptable.
3. Intraocular pressure ≥ 36mmHg (unmedicated) in either eye (individuals who are excluded for this criterion are not allowed to attempt requalification), or use of more than two ocular hypotensive medications within 30 days of screening. Note: fixed dose combination medications, for the purpose of this exclusion criterion, count as one medication. However, subjects currently taking 2 fixed dose combination products are excluded.
4. Treatment-naïve subjects.
5. Prior treatment with GANFORT® topical eye drops where the subjects IOP did not achieve the target IOP and was considered either a therapeutic failure or to have insufficient response. Subjects currently (immediately prior to screening visit) being treated with GANFORT® are excluded from the study.
6. Known hypersensitivity to any component of the investigational formulations to be used (e.g., benzalkonium chloride) or to fluorescein.
7. Previous glaucoma intraocular surgery, including SLT or ALT in either eye.
8. Refractive surgery in either eye (e.g., radial keratotomy, PRK, LASIK, corneal cross-linking, keratoplasty).
9. Ocular trauma within the six months prior to screening, or ocular surgery or non-refractive laser treatment within the three months prior to screening.
10. Recent or current evidence of ocular infection or inflammation in either eye. Current evidence of clinically significant blepharitis, conjunctivitis, keratitis, current evidence or history of herpes simplex or zoster keratitis in either eye at screening.
11. Use of ocular medication in either eye of any kind within 30 days of screening and throughout the study, with the exception of a) ocular hypotensive medications which must have been the same medication for 30 days prior to screening (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after, screening), c) lubricating drops for dry eye (which may be used throughout the study), as prescribed by the Investigator.
12. Mean central corneal thickness greater than 620μm at screening.
13. Any abnormality preventing reliable Goldmann applanation tonometry of either eye (e.g., keratoconus).

    Systemic:
14. Clinically significant abnormalities in laboratory tests at screening.
15. Known hypersensitivity or contraindication to GANFORT® (Appendix 3 Marketed Product Medication Information Section 4.3) and to β-adrenoceptor antagonists (e.g. Chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure or heart rate; second or third-degree heart block or congestive heart failure, cardiac failure, cardiac shock and severe diabetes).
16. Clinically significant systemic disease which might interfere with the study.
17. Participation in any investigational study within 30 days prior to screening.
18. Systemic medication including corticosteroid containing drugs that could have a substantial effect on IOP which HAVE NOT been maintained at a consistent dose and regime within 30 days prior to screening, and are anticipated to change in dose and/or regime during the study.
19. Use of topical steroid containing medications on the face or in or around the eyes will exclude the subject (see Section 5.6 Concomitant Medications).
20. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable and highly effective form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal (1 year without menses with appropriate clinical profile, e.g. age appropriate, > 45 years in the absence of HRT. In questionable cases the subject must have FSH value > 40mIU/mL and an estradiol value < 40pg/mL (< 140pmol/L)) or three months post-surgical sterilization.
21. Vulnerable subjects such as minors, adults under legal protection or unable to express their consent (e.g. hospitalized persons in coma), persons deprived of liberty (prisoners from jails), or persons subject to psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Study Director — Aerie Pharmaceuticals Inc.
Locations (68):
- Austria (3):
  - State Hospital - University Medical Center Academical Department of Ophthalmology, Graz
  - Albertgasse 39/10+11, Vienna
  - Hanusch Hospital, Vienna
- UZ Leuven, campus Gasthuisberg, Herestraat 49, 3000 Leuven, Leuven, Belgium
- Czechia (2):
  - Faculty Hospital Brno Eye Department, Brno
  - Glaucoma center Oční klinika VFN a 1. LF UK, Prague
- France (5):
  - Ophthalmology Service Centre Francois Xavier Michelet CHU Pellegrin, Bordeaux
  - Centre ophtalmologique Pole vision val d'ouest, Écully
  - Ophthalmology Service - Batiment R Hospital de la Croix-Rousse, Lyon
  - CHU de Nantes-Hospital Hotel Dieu Ophthalmology Service, Nantes
  - Ophthalmology department Necker University Hospital-Enfants Malades, Paris
- Germany (5):
  - University Medical Center Freiburg, Eye Center,Killianstr.5, Freiburg i. Breisgau, Freiburg im Breisgau
  - Department of Ophthalmology Clinical Johannes Gutenberg-University Mainz, Mainz
  - Universitats-Augenklinik, Studienzentrum/Clinical Trials in Opthalmology (CTO), Münster
  - University Eye Hospital Tuebingen, STC eyetrial at the center for Ophthalmolgy, Tübingen
  - Augenarztpraxis Dr. Andreas Bayer, Weilheim
- Hungary (7):
  - Budapest Retina Associates, Budapest
  - Department of Ophthalmology Semmelweis University, Budapest
  - University of Debrecen, Clinical Center, Ophthalmology Department, Debrecen
  - Clinexpert Gyongyos Kft., Heves
  - Ganglion Medical Center, Pécs
  - University of Szeged, Department of Ophthalmology, Szeged
  - Markusovszky University Teaching Hospital, Szombathely
- Italy (12):
  - Ophthalmic Clinic DiNOGMI University Hospital San Martino, Genova
  - ASST Fatebenefratelli Sacco P.O.L.Sacco, Milan
  - ASST Santi Paolo e Carlo - Ophthalmic Clinic, Milan
  - Dept. Ophthalmology, San Raffaele Hospital, Milan
  - Department of Medicine and Surgery University of Parma, Parma
  - Ophthamic Clinic of the University of Pavia, IRCCS Foundation San Matteo Policlinic, Pavia
  - AOU Pisana Hospital of Cisanello, Pisa
  - G.B.Bietti Foundation - IRCCS, Rome
  - Senese University Hospital, Siena
  - S.C.U Oculistica, Azienda Ospedaliero Universitaria, Città della Salute e della Scienza, Torino
  - University Eye Clinic Ospedale Maggiore, Trieste
  - Politecnico Gianbattista Rossi AOUI Ospedale Borgo Roma, Verona
- Latvia (4):
  - Signes Ozolinas Doctor Practice in Ophthalmology, Jelgava
  - Latvian American Eye Centre (LAAC), Riga
  - P.Stradins Clinical University Hospital, Ophthalmology Clinic, Riga
  - Riga East University hospital, In-patient Department "Biķernieki", Ophthalmology Clinic, Riga
- Poland (4):
  - Professor K. Gibinski University Clinical Centre, Katowice
  - Ophthalmic Clinic Jasne Blonia, Lodz
  - Department of Diagnostics and Microsurgery of Glaucoma, Lublin
  - Military Institute of Medicine Klinika Okulistyki, Warsaw
- Spain (13):
  - Centro de Ojos de la Coruña, A Coruña
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital General de Catalunya Ophthalmology Department, Barcelona
  - Hospital QuironSalud Barcelona, Barcelona
  - Institut Catala de retina (ICR) Glaucoma and Investigation Department, Barcelona
  - Hospital General del S.A.S. de Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofía de Córdoba, Córdoba
  - Hospital Universitario Virgen Macarena Ophthalmology Department, Seville
  - Hospital Universitario de Torrevieja Ophthalmology Department, Torrevieja
  - FISABIO-Oftalmología Médica, Valencia
  - Ophthalmology Department Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa Zaragoza Ophthalmology department, Zaragoza
  - Hospital Universitario Miguel Servet Ophthalmology Department, Zaragoza
- United Kingdom (12):
  - City Hospitals Sunderland NHS Foundation Trust Sunderland Eye Infirmary, Sunderland, Tyne and Wear
  - NHS Grampian Aberdeen Royal Infirmary, Aberdeen
  - Cambridge University Hospitals NHS Trust, Cambridge
  - Ophthalmology Department, Queen Alexandra Hospital, Cosham
  - Mid-Cheshire Hospitals NHS Foundation Trust, Crewe
  - Northwest Anglia NHS Foundation trust Hinchingbrooke Hospital, Huntingdon
  - Guy's & St Thomas' NHS Foundation Trust Glaucoma Research Area, London
  - King's College Hospital, London
  - Moorfields Eye Hospital NHS, London
  - Western Eye Hospital, London
  - Royal Hallamshire Hospital, Sheffield
  - Queen Mary Hospital, King's College Hospital NHS, Sidcup

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in 11 European countries between September 2017 and May 2020.
Pre-assignment Details: All participants underwent a period of washout for their pre-study ocular hypotensive medication for a prescribed period (up to 4 weeks or longer), depending on the medication, before receiving study medication.
  From the total 436 participants, 6 were not included in the analysis due to serious GCP breaches (2 from the Netarsudil/Latanoprost 0.02%/0.005% arm and 4 from the Ganfort arm).
  The remaining 430 participants (218 and 212 respectively) were included in the analysis.
Period: Overall Study
Arm/Group | Netarsudil/Latanoprost 0.02%/0.005% | GANFORT®
Started | 218 | 212
Intent-to-Treat Population (All randomized participants who received at least one dose of study medication.) | 218 | 212
Per-Protocol Population (Subset of the ITT Population, includes participants (and their visits) who did not have major protocol violations likely to seriously affect the primary outcome of the study as judged by a masked evaluation prior to the unmasking of the study treatment.) | 169 | 170
Safety Population (All randomized participants who received at least one dose of study medication.) | 218 | 212
Completed | 163 | 199
Not Completed | 55 | 13
Not completed — Adverse Event | 40 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Disallowed Concurrent Medication | 1 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Death | 0 | 1
Not completed — Other - Reason not reported in CSR | 4 | 3

BASELINE CHARACTERISTICS:
Population: 436 participants were randomized; 220 to the Netarsudil/Latanoprost 0.02%/0.005% arm and 216 to the Ganfort arm.
  From the total 436 participants, 6 were not included in the analysis due to serious GCP breaches (see Pre-Assignment Details for more information).
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil/Latanoprost 0.02%/0.005% | GANFORT® | Total
Number analyzed (Participants) | 218 | 212 | 430
Age, Categorical [Count of Participants; unit: Participants] — Participants were randomized on a 1:1 ratio to either group. Age was not a consideration for group assignment.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 71 | 79 | 150
    >=65 years | 147 | 133 | 280
Age, Continuous [Mean (Full Range); unit: years] — Participants were randomized on a 1:1 ratio to either group. Age was not a consideration for group assignment.
  years
    Mean | 67.3 [25 to 91] | 67.0 [22 to 91] | 67.2 [22 to 91]
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were randomized on a 1:1 ratio to either group. Gender was not a consideration for group assignment.
  Participants
    Female | 131 | 92 | 223
    Male | 87 | 120 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 56 | 117
  Not Hispanic or Latino | 157 | 156 | 313
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 210 | 200 | 410
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Austria | 17 | 17 | 34
  Latvia | 8 | 8 | 16
  Belgium | 5 | 5 | 10
  Hungary | 8 | 11 | 19
  Czechia | 30 | 31 | 61
  Poland | 3 | 3 | 6
  Italy | 21 | 21 | 42
  United Kingdom | 20 | 15 | 35
  France | 2 | 4 | 6
  Germany | 38 | 36 | 74
  Spain | 66 | 61 | 127

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal Intraocular Pressure by Goldmann Applanation Tonometry
Description: Comparison of PG324 to Ganfort for mean intraocular pressure at specified timepoints at Week 2, Week 6 and Month 3.
Time Frame: Day 90
Population: A total of 430 (100%) participants were included in the Safety and Intent-to-Treat populations.
Measure: Least Squares Mean (Full Range); unit: mmHg
Arm/Group | Netarsudil/Latanoprost 0.02%/0.005% | GANFORT®
Number analyzed (Participants) | 218 | 212
mmHg
  Week 2 | 15.39 [15.09 to 15.84] | 15.56 [15.42 to 15.67]
  Week 6 | 15.64 [15.18 to 16.20] | 15.25 [15.16 to 15.32]
  Month 3 | 15.61 [15.28 to 15.93] | 15.19 [15.09 to 15.27]
Statistical Analysis 1: Comparison: Netarsudil/Latanoprost 0.02%/0.005% vs GANFORT®; Assuming no difference between PG324 and Ganfort, a two-tailed alpha of 0.05 (2-sided 95% CI) at each of 9 time points, a common SD of 3.5 mmHg, and a correlation between time points of ≤ 0.60, 200 ITT subjects per arm were necessary to have 85% power to show clinical non-inferiority of PG324 to Ganfort in the mean change from baseline IOP; Test type: Other — The primary analysis was performed on the ITT population with imputation by Markov Chain Monte Carlo method; p < 0.05, Regression, Linear — Linear model with IOP at the given visit and time point as the response, baseline IOP as a covariate, and treatment as a main effect factor at each time point (08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 Visits); Non-inferiority for PG324 was concluded if the UL of the 95% CI was ≤ l.5 mmHg at all 9 time points and ≤ l.0 mmHg at the majority of time points

ADVERSE EVENTS:
Time Frame: Adverse events were documented for each participant from the time of signing consent until 30 days after the last dose of Investigational Product. This was a maximum period of approximately 9 months (38 weeks) for participants who completed the full study duration.
Arm/Group | Netarsudil/Latanoprost 0.02%/0.005% | GANFORT®
All-Cause Mortality (participants affected / at risk) | 0/218 | 1/212
Serious Adverse Events (participants affected / at risk) | 7/218 | 7/212
Other Adverse Events (participants affected / at risk) | 117/218 | 53/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Netarsudil/Latanoprost 0.02%/0.005% (N=218) | GANFORT® (N=212)
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Ischemic stroke (Nervous system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil/Latanoprost 0.02%/0.005% (N=218) | GANFORT® (N=212)
Conjunctival Hyperemia (Eye disorders) | 72 (72) | 23 (23)
Cornea Verticillata (Eye disorders) | 24 (24) | 0 (0)
Conjunctival Hemorrhage (Eye disorders) | 18 (18) | 5 (5)
Eye Pruritus (Eye disorders) | 17 (17) | 4 (4)
Punctate Keratitis (Eye disorders) | 12 (12) | 5 (5)
Conjunctivitis Allergic (Eye disorders) | 12 (12) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 11 (11) | 10 (10)
Hypertension (Vascular disorders) | 10 (10) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03284853/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03284853/SAP_001.pdf